CLINICAL TRIAL: NCT00222963
Title: Pilot Study to Assess the Effectiveness of Tonsil and Adenoidectomy (T+A) in Overweight Children and Adolescents
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: HV Connolly, MD, U of R
Other Study IDs: 10297
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2006-09

CONDITIONS: Obesity; Obstructive Sleep Apnea Syndrome
Keywords: Obesity; Obstructive Sleep Apnea Syndrome; Children; Adolescents; Adenotonsillectomy
MeSH Terms: conditions — Obesity; Sleep Apnea, Obstructive

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Obesity has reached epidemic proportions in the United States with roughly 20% of American children being overweight and has serious consequences such as sleep apnea.Additionally, obesity is known to result in the earlier onset of puberty . Thus, it can be expected that obese children take-on adult characteristics at an earlier chronologic age than their non-obese counterparts. Current guidelines recommend adenotonsillectomy (T+A) as primary and effective therapy for sleep apnea resulting in polysomnographic resolution in 75-100% of patients. Small studies have shown that T+A relieves symptoms in obese children but surgical intervention has been less efficacious in adults. We hypothesize that T+A may be less efficacious in obese adolescents because of earlier onset of puberty imparting more adult characteristics. We further hypothesize that the efficacy of T+A will correlate more closely with Tanner staging than with chronologic age because of the earlier onset of sexual maturation associated with obesity.

DETAILED DESCRIPTION:
Obesity has reached epidemic proportions in the United States with roughly 20% of American children being overweight . Obesity has serious health consequences increasing the risk of hypertension , type II diabetes and obstructive sleep apnea . Additionally, obesity is known to result in the earlier onset of puberty . Thus, it can be expected that obese children take-on adult characteristics at an earlier chronologic age than their non-obese counterparts.

Similarly, sleep apnea is a common problem with wide reaching consequences including increased risk for hypertension , insulin resistance and neurocognitive dysfunction leading to poor academic performance . Furthermore, sleep fragmentation produced by repetitive episodes of nocturnal apnea may lead to daytime somnolence and increased food intake as a behavioral attempt to overcome sleepiness and thereby further contribute to obesity .

Current guidelines recommend adenotonsillectomy (T+A) as primary and effective therapy for sleep apnea resulting in polysomnographic resolution in 75-100% of patients. Small studies have shown that T+A relieves symptoms in obese children but surgical intervention has been less efficacious in adults . Although nocturnal polysomnogrpahy (NPSG) is considered the gold standard by which to diagnose obstructive sleep apnea (OSAS), published studies assessing the efficacy of treatment in obese children using polysomngraphy to objectively quantify the degree of sleep apnea before and after T+A do not exist.

Surgical intervention may not be indicated in children without adenotonsillar hypertrophy. Similarly, children who are at high risk for surgical or anesthetic related complications may be deemed poor surgical candidates. For these children as well as those who fail T+A, non-invasive, continuous positive airway pressure (CPAP) applied via a nasal mask is effective in treating sleep disordered breathing. However, CPAP is effective only when in use and multiple studies demonstrate low rates of long-term compliance in adults . No studies assessing children's adherence with CPAP exist. Certainly, it is expected that compliance in the adolescent population would be similar, if not worse than adults. Thus, CPAP is not recommended as first-line therapy when surgical intervention is viable.

We hypothesize that T+A may be less efficacious in obese adolescents because of earlier onset of puberty imparting more adult characteristics. We further hypothesize that the efficacy of T+A will correlate more closely with Tanner staging than with chronologic age because of the earlier onset of sexual maturation associated with obesity. Thus, we propose to study the efficacy of T+A in the treatment of sleep apnea in obese adolescents using polysomnography to quantify the severity of OSAS before and after T+A. It is anticipated that results from this preliminary study will be used to form the basis for studies comparing efficacy of adenotonsillectomy against the use of CPAP in this population.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8-18 who are overweight or at risk for overweight (defined as BMI >85%ile for age and gender referred for evaluation and treatment of sleep apnea.

Exclusion Criteria:

* Children with underlying craniofacial anomalies, chromosomal abnormalities, neuromuscular disorders and metabolic disorders except diabetes will be excluded. Children and parents who do not speak or write English will be excluded. Children with neuropsychiatric disabilities severe enough to preclude sufficient cooperation with overnight polysomnography will also be excluded.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 250 (Actual)
Dates: Start 2004-09

CONTACTS AND LOCATIONS:
Overall Officials: Heidi V. Connolly, MD, Principal Investigator — University of Rochester; Margaret-Ann Carno, PhD,RN, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States